CLINICAL TRIAL: NCT00760448
Title: Trial Investigating the Hypoglycaemic Response to Single Doses of Insulin Detemir and NPH Insulin in Subjects With Type 1 Diabetes
Brief Title: Comparison of Insulin Detemir and NPH With Respect to Lowering the Blood Sugar and Symptoms Experienced by Type 1 Diabetics During Hypoglycaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1449
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in UK. The aim of this clinical trial is to investigate lowering the blood sugar and symptoms experienced during hypoglycaemia

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities.
* Type 1 diabetes
* Treatment with insulin for minimum three months
* Duration of diabetes for more than 12 months
* Body Mass Index (BMI) less than 30 kg/m2
* HbA1c equal to or greater than 10 % based on analysis from central laboratory

Exclusion Criteria:

* Participation in any other clinical trial involving other investigational products within the last three months
* Current treatment with insulin in a daily dose above 100 U
* Episode of symptomatic hypoglycaemia, or a capillary plasma glucose value of less than 3.5 mmol/L in the past two weeks
* Hypoglycaemic unawareness or severe autonomic neuropathy
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers and MAO inhibitors
* Current treatment with oral antidiabetic drugs
* Impaired hepatic function measured as ALAT of more than two times the upper reference limit
* Impaired renal function measured as creatinine of more than 150 micromol/L (1.7 mg/dL)
* Cardiac problems defined as decompensated heart failure (NYHA class III and IV) at any time and/or angina pectoris and/or myocardial infarction within the last 12 months
* Known or suspected allergy to trial product or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Blood donation of more than 500 mL within the last three months
* Any condition that the Investigator and/or the Sponsor feels would interfere with study participation or evaluation of results
* Pregnancy or intention of becoming pregnant, breast-feeding or judged to be using inadequate contraceptive methods. Adequate contraceptive methods are sterilisation, intrauterine device (IUD), oral contraceptives or consistent use of barrier methods
* Previous participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted hypoglycaemic symptoms score at nadir plasma glucose concentration based on the Edinburgh Hypoglycaemia Scale: autonomic symptoms, neuroglycopenic symptoms and general malaise | From -40 min and until immediately before trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Guildford, United Kingdom

REFERENCES:
- [Result] Smeeton F, Shoajee-Moradie F, Jackson N, Westergaard L, Endahl L, Haahr HL, Umpleby M, Russell-Jones D. No Difference in Cognitive Function, Symptons or Counter-regulatory Responses after Induced Hypoglycemia in Subjects with Type 1 Diabetes. ADA 2007 2007; 56 (Suppl. 1): A168 (634-P)
- [Derived] Smeeton F, Shojaee Moradie F, Jones RH, Westergaard L, Haahr H, Umpleby AM, Russell-Jones DL. Differential effects of insulin detemir and neutral protamine Hagedorn (NPH) insulin on hepatic glucose production and peripheral glucose uptake during hypoglycaemia in type 1 diabetes. Diabetologia. 2009 Nov;52(11):2317-23. doi: 10.1007/s00125-009-1487-4. Epub 2009 Aug 26. PMID 19707744
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com